CLINICAL TRIAL: NCT03525262
Title: A Phase II Randomized Controlled Trial of Stereotactic Ablative Body Radiotherapy (SAbR) With or Without Neurovascular Sparing for Erectile Function Preservation in Localized Prostate Cancer
Brief Title: Prostate Oncologic Therapy While Ensuring Neurovascular Conservation (POTEN-C)
Acronym: POTEN-C
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Neil Desai, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 092017-018
Record Dates: First submitted 2018-04-23; First posted 2018-05-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer Adenocarcinoma
Keywords: Erectile dysfunction, Neurovascular, Prostate, Rectal spacer, Radiotherapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAbR WITHOUT Neurovascular sparing (No Intervention): * GTV represents MR defined dominant radiographic disease, if identifiable.
  * CTV encompasses the full prostate. At physician's discretion, the insertion of the seminal vesicle upon the prostate on slices containing prostate may be included.
  * PTV1_30Gy will not be used or created on this arm
  * PTV2_SAbR40Gy OR PTV2_SAbR45Gy will be generated by a 3mm expansion on the CTV. PTV2_SAbR will receive 8-9 Gy per fraction for 5 fractions (40-45 Gy).
- SAbR WITH Neurovascular sparing (Experimental): * GTV represents MR defined dominant radiographic disease, if identifiable.
  * CTV encompasses the full prostate. At physician's discretion, the insertion of the seminal vesicle upon the prostate on slices containing prostate may be included.
  * PTV1_30Gy represents a 3mm expansion on the CTV, excluding the neurovascular structures on the side to be spared (left or right). PTV1 will receive 6 Gy per fraction for 5 fractions (30 Gy).
  * PTV2_SAbR40Gy OR PTV2_SAbR45Gy will be generated by subtracting a 5mm expansion around the neurovascular elements to be spared (at least one side, left or right) from PTV1. These neurovascular structures consist of the neurovascular bundle, penile bulb, and internal pudendal arteries (see 4.1.5.2.16). PTV2 will receive 8-9 Gy per fraction for 5 fractions (40-45 Gy).
  Interventions: Radiation: 30Gy (Gray) planning target volume (PTV)

INTERVENTIONS:
Radiation: 30Gy (Gray) planning target volume (PTV) — PTV1_30Gy represents a 3mm expansion on the prostate (and proximal seminal vesicle per physician discretion), excluding the neurovascular structures on the side to be spared (left or right). PTV1 will receive 6 Gy per fraction for 5 fractions (30 Gy).
  Arms: SAbR WITH Neurovascular sparing

SUMMARY:
Reduction of dose to or 'sparing' of neurovascular structures during stereotactic ablative body radiotherapy (SAbR) for localized prostate cancer will improve retention of sexual potency, while retaining excellent oncologic control and other secondary health-related quality of life (HRQOL) endpoints.

Primary Objectives:

• To compare the decline in patient health-related quality of life (HRQOL) instrument-defined erectile dysfunction following stereotactic ablative body radiotherapy (SAbR) with or without neurovascular sparing

Secondary Objectives:

* Assess acute (within 3 months of treatment) and chronic (>3 months after treatment) SAbR related GU and GI toxicities, as well as serial impact on HRQOL metrics over time
* Assess biochemical progression free survival, local recurrence, distant recurrence, and survival
* Evaluate simplified 'practical' secondary HRQOL sexual potency endpoints that can be compared to prior literature.

Exploratory Objectives:

* Evaluate feasibility of MRI BOLD/TOLD to be integrated as hypoxia monitoring sequences to standard already planned diagnostic and/or treatment planning MRI on the study in five patient pilot.
* Evaluate quality of spacer placement and its effect on dose to neurovascular structures
* Evaluate rate local recurrence in the area of sparing adjacent to the neurovascular elements by biopsy in those with biochemical progression.

DETAILED DESCRIPTION:
This is a phase II randomized, multi-institution, open-label, patient and HRQOL endpoint assessor blinded study evaluating the ability of neurovascular element sparing SAbR to decrease erectile dysfunction. The study procedure is to reduce 2-year Expanded prostate cancer index composite (EPIC) sexual domain score decline by 50% (-20 to -10), there by improving potency preservation. This reduction is usually expected to observe in patients undergoing the treatment stereotactic ablative body radiotherapy (SAbR) to 40-45 Gy with rectal spacer +/- sparing of at least one side's neurovascular structures using dose-painting.

Primary Endpoint:

• The Expanded prostate cancer index composite (EPIC) health-related quality of life (HRQOL) instrument includes a sexual function domain, which is used to produce a composite score of 0-100 from 9 questions related to ability to achieve an erection with or without aids and participate in intercourse. The primary endpoint will be the mean 24-month decline in EPIC sexual function domain composite score.

Secondary Endpoints:

* Acute Genitourinary (GU) and Gastrointestinal (GI) toxicity is defined as grade 1-5 toxicity occurring prior to 270 days from the start of protocol treatment. It is graded based on CTCAE v4.0.
* Delayed GU and GI toxicity is defined as grade 1-5 toxicity occurring prior to 270 days from the start of protocol treatment. It is graded based on CTCAE v4.0.
* Non GU and GI toxicity up to six months post treatment.
* Biochemical failure Radiation therapy oncology group-American Society for Therapeutic Radiology and Oncology (RTOG-ASTRO) definition (also known as Phoenix definition) - Thus, when the Prostate Specific Antigen (PSA) rises by more than 2 ng/ml above the lowest level (nadir) achieved after treatment, biochemical failure has occurred and the date of the failure is recorded at the time the nadir plus 2 ng/ml level is reached. Patients should be followed for a minimum of 5 years on this study to evaluate this endpoint.
* Overall survival
* Disease-specific survival
* Clinical progression including local/regional and distant relapse
* HRQOL questionnaires (EPIC and SF-12)
* Erectile function medication and device aids tracked before and after therapy longitudinally
* Feasibility of MRI BOLD/TOLD in evaluating tumor hypoxia in no more than five patient pilot

Sample Size: To enroll 120 patients (60 patients in each treatment arm).

The sample size is estimated, first, assuming that neurovascular element sparing SAbR (experimental arm intervention) will result in a mean 24 month decline in EPIC (HRQOL instrument) sexual domain composite score of -20, as compared to a decline of -10 in a standard SAbR without neurovascular element sparing. A total sample size of 102 patients (51 patients in each treatment group) achieves 80% power to detect this difference of 10 in EPIC sexual domain composite score decline at 24 months after treatment, with an equal standard deviation of 20 in both groups and at a two-sided significance level of 0.10, using a two-sample t-test (effect size 0.50).

An attrition rate of EPIC sexual domain questionnaire completion at 2-years of 15% is anticipated, based upon yields from multi-center prospective trials in prostate cancer radiotherapy with EPIC HRQOL endpoints. A total of 120 patients will be accrued to account for this 15% attrition rate.

Statistical Analysis: For the primary endpoint, a two-sided two-sample t-test will be used to compare EPIC sexual function domain score composite declines at 24 months from treatment between experimental SAbR arms with and without neurovascular sparing. Our sample size of 60 patients in each arm gives a calculated 80% power to detect a difference of 10 (considered the minimally important difference for sexual domain) at a two-sided significance level 0.10, assuming an equal standard deviation of 20 in both groups and allowing for 15% attrition in survey completion. Secondary endpoints and their analysis methodology is further specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Appropriate staging studies identifying patient as AJCC 7th edition clinical stage T1 (a, b, or c) or T2 (a, b, or c) adenocarcinoma of the prostate gland. The patient should not have direct evidence of regional or distant metastases after appropriate staging studies. See Appendix I for details on AJCC 7th Edition staging criteria. Histologic confirmation of cancer will be required by biopsy performed within 12 months of registration. T-staging may be assessed by multi-parametric imaging alone if digital rectal examination was deferred.
3. The patient's Zubrod performance status must be 0-2 (see Appendix II for definition).
4. The Gleason summary score should be less than or equal to 7 [Grade group 1 (Gleason 3+3=6), group 2 (Gleason 3+4=7), and group 3 (Gleason 4+3=7) are allowed]. See Appendix III for details on definitions. While a template biopsy is recommended, it is not required in the case of MRI fusion biopsy performed on all dominant MR lesions (defined as PIRADS v2 4-5).
5. Baseline AUA symptom score ≤19 (see Appendix IV for questionnaire) without need for maximum medical therapy (specifically, not on tamsulosin 0.8mg daily).
6. EPIC sexual domain composite score 60-100 (see Appendix V).
7. Multi-parametric MRI evaluation of the prostate is required for this study within 12 months of registration. Gross radiographic disease on MRI (defined as PIRADS v2 score 3-5) must be > 5mm at minimum distance from at least one side's neurovascular bundle, which is typically the closest of the neurovascular elements to the prostate.
8. The serum PSA should be less than or equal to 20 ng/ml within 90 days of registration.

   -Study entry PSA must not be obtained during the following time frames: (1) 10-day period following prostate biopsy; (2) following initiation of ADT or anti-androgen therapy; (3) within 30 days after discontinuation of finasteride; (4) within 90 days after discontinuation of dutasteride; (5) within 5 days of a digital rectal examination (which is not a required exam on the protocol).
9. Ultrasound or MRI based volume estimation of prostate gland ≤ 80 grams. Cytoreduction therapy (finasteride or dutasteride only) may be considered for those with >60 gram size.
10. All patients must be willing and capable to provide informed consent to participate in the protocol within the 30 days prior to registration.

Exclusion Criteria:

1. Subjects with clinical (digital rectal examination) evidence of extraprostatic extension (T3a) or seminal vesicle involvement (T3b). MRI evidence of equivocal/potential but not definite extraprostatic extension is allowed, as long as it is unilateral and not on the side of the gland proposed for neurovascular element sparing. In equivocal cases of potential extracapsular extension on MRI only, discretion is left to the treating physician.
2. MRI evidence of gross disease (defined as PIRADS v2 score 3-5 lesions) ≤5mm of BOTH neurovascular bundles, which are the most proximate of the neurovascular elements planned for sparing on this protocol.
3. Patients with all three intermediate risk factors (PSA >10 and ≤ 20, Gleason 7, clinical stage T2b-T2c) who ALSO have ≥50% of the number of their template biopsy cores positive for cancer are ineligible.
4. Inability to undergo multi-parametric MRI.
5. Evidence of metastatic disease. Note bone scan is not required for this study given the low-intermediate NCCN risk cohort to be enrolled.
6. Evidence of clinical nodal involvement of the pelvis. Biopsy is required for lymph nodes over ≥1.5cm in short-axis measured size.
7. No currently active ADT or anti-androgen therapy at time of registration is allowed. Further, no more than 3 cumulative months of prior ADT or anti-androgen therapy is allowed. If either has been used by the patient, there must be a demonstration of testosterone recovery (>50ng/dL serum blood level), EPIC sexual domain score ≥60, and at least 1 month between demonstration of testosterone recovery and study registration (any one measurement of testosterone recovery suffices).
8. Testosterone ≤ 50 ng/dL (any one measurement >50 ng/dL suffices for inclusion) within 90 days of study entry.
9. Subjects who have had previous pelvic radiotherapy or have had chemotherapy or surgery for prostate cancer.
10. Subjects who have plans to receive other concomitant or post treatment adjuvant antineoplastic therapy while on this protocol including surgery, cryotherapy, conventionally fractionated radiotherapy, hormonal therapy, or chemotherapy given as part of the treatment of prostate cancer.
11. Subjects who have undergone previous transurethral resection of the prostate (TURP) within 1 year of enrollment or ablative procedures to the prostate for benign prostatic hyperplasia or other conditions (i.e. cryotherapy, HIFU).
12. Subjects who have baseline severe urinary symptoms, as defined by AUA symptom score >19 (alpha-blocker medication allowed except if taking tamsulosin 0.8mg daily at baseline which indicates compensated severe symptoms and also can affect sexual function).
13. Subjects who have a history of significant psychiatric illness that would confound informed consent.
14. Severe, active co-morbidity, defined as follows:

    1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
    2. Myocardial infarction within the last 6 months
    3. Acute bacterial or fungal infection requiring intravenous antibiotics at time of registration
    4. Patients with active inflammatory colitis (including Crohn's Disease and ulcerative colitis) currently requiring systemic steroids and/or systemic immunosuppression are not eligible.
15. Subjects with a known allergy to polyethylene glycol hydrogel (rectal spacer material) or contraindication to spacer products (SpaceOAR).
16. Subjects with uncontrolled coagulation disorder which cannot be controlled with anticoagulants.
17. Men active with partners of reproductive potential who do not agree that they will use an effective contraceptive method during treatment and 6 months after treatment.
18. Men who require erectile function medication or aid to achieve an erection sufficient for intercourse. Ability to achieve erection sufficient for intercourse without medication or aid at least once time in the month prior to registration is sufficient for inclusion.
19. Men who have clinically significant penile malformation (i.e. Peyronie's disease) or history of penile implantation are excluded.
20. If DRE is performed, patient may not have palpable disease on side of gland to be planned for neurovascular sparing. Given the poor accuracy of DRE, such a finding should be confirmed by MRI and/or biopsy to harbor actual disease before excluding a patient on this basis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
To compare the decline in patient health-related quality of life. | Mean 24-Months
  To compare the decline in patient health-related quality of life (HRQOL) instrument-defined erectile dysfunction following stereotactic ablative body radiotherapy (SAbR) with or without neurovascular sparing. The Expanded Prostate Cancer Index Composite (EPIC) health-related quality of life (HRQOL) instrument includes four sub-scales like urinary function, bowel habits, sexual function, and hormonal function. The primary outcome (sexual function) which has a range score of 0-100 from 9 questions related to ability to achieve an erection with or without aids and participate in intercourse. Higher the score represents the better outcome. Individual responses are summed for a total score of sexual function.

SECONDARY OUTCOMES:
Acute & Chronic Genitourinary (GU) and Gastrointestinal (GI) toxicity | Mean 24-Months
  Assess acute (within 3 months of treatment) and chronic (>3 months after treatment) SAbR related GU and GI toxicities, as well as serial impact on HRQOL metrics over time. Severity or Toxicity will be assessed according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. The consequences of gastointestinal/renal/genitourinary/sexual and reproductive toxicity should all be graded 1-5 according to the Common Terminology Criteria For Adverse Events (CTCAE), version 4.0 occurring prior to 270 days from the start of protocol treatment. Other treatment related toxicity attributed to the therapy will be captured, recorded and the consequences of should all be graded 1-5 according to the Common Terminology Criteria For Adverse Events (CTCAE). CTCAE V4.0 along with grades 1-5 is provided in the link for reference (https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03/CTCAE_4.03_2010-06-14_QuickReference_8.5x11.pdf).
Biochemical progression free survival. | 60 Months
  Assess biochemical progression free survival. Biochemical failure RTOG-ASTRO definition - when the PSA rises by more than 2 ng/ml above the lowest level (nadir) achieved after treatment, biochemical failure has occurred and the date of the failure is recorded at the time the nadir plus 2 ng/ml level is reached.
Time to local recurrence. | 60 Months
  The time to progression will be measured from the date of study entry to the date of documented local progression as determined by clinical exam and/or MRI. Local progression is defined by progression within the prostate, seminal vesicles or immediately adjacent extracapsular soft tissue. Biopsy confirmation is not required but is encouraged.
Time to distant recurrence. | 60 Months
  The time to distant failure will be measured from the date of study entry to the date of documented regional nodal recurrence or distant disease relapse. Patients with evidence of biochemical failure, but a negative prostate biopsy, will be considered as distant failure only.
Overall survival. | 60 Months
  The survival time will be measured from the date of accession to the date of death. All patients will be followed for survival. Every effort should be made to document the cause of death.
Evaluate simplified 'practical' secondary HRQOL sexual potency endpoints. | Mean 24-Months
  Evaluate simplified 'practical' secondary HRQOL sexual potency endpoints that can be compared to prior literature. The Expanded Prostate Cancer Index Composite (EPIC) health-related quality of life (HRQOL) instrument includes four sub-scales like urinary function, bowel habits, sexual function, and hormonal function. The primary outcome (sexual function) which has a range score of 0-100 from 9 questions related to ability to achieve an erection with or without aids and participate in intercourse. Higher the score represents the better outcome. Individual responses are summed for a total score of sexual function.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCSF ( Department of Radiation Oncology University of California San Francisco), San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Penrose Hospital, Colorado Springs, Colorado
  - University of Michigan- Michigan Medicine, Ann Arbor, Michigan
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Penn Medicine Radiation Oncology, Philadelphia, Pennsylvania
  - UT Southwestern Cancer Center, Dallas, Texas